CLINICAL TRIAL: NCT04250766
Title: Diagnostic Performances of Preoperative Echo-guided Uterine Biopsy in the Management of Suspect Uterine Sarcoma Tumors
Brief Title: Diagnostic Performances of Preoperative Echo-guided Uterine Biopsy in the Management of Suspect Uterine Sarcoma Tumors (BIOPSAR)
Acronym: BIOPSAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: GIRCI SOHO (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IB 2018-02; 2018-A02343-52 (Other: ID-RCB number)
Record Dates: First submitted 2019-11-15; First posted 2020-01-31 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Fibroid Uterus; Sarcoma Uterus
Keywords: Uterine fibroma; Suspect uterine sarcoma; Echo-guided biopsy
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm echo-guided uterine biopsy (Other)
  Interventions: Procedure: Echo-guided uterine biopsy

INTERVENTIONS:
Procedure: Echo-guided uterine biopsy — Echo-guided uterine biopsy will be performed by a specialized radiologist by transvaginal and exclusive transuterine approach. 4 to 5 samples will be made.
  Local anesthesia will be performed. A pain assessment will be performed during the biopsy (visual or verbal scale).

SUMMARY:
This is a prospective multi-center interventional study that will be performed in an effort to assess the diagnostic accuracy performance of preoperative vaginal ultrasound-guided biopsy (VUGB) to detect the exact histology of uterine tumors and thereafter triage cases being eligible for morcellation during laparoscopic resection. Ten tertiary French centers will participate in the present study.

DETAILED DESCRIPTION:
Prior to carrying out the research, the informed consent of the person must be obtained after being informed of the purpose of the research, its conduct and duration, benefits, potential risks and constraints of the study.

During the inclusion check-up, exams must be performed within 30 days before the guided echo biopsy: clinical examination, gynecological examination, pain assessment (visual or verbal scale), biological and radiological assessment (Doppler ultrasound Pelvis and MRI pelvis).

The echo-guided biopsy will be performed by a specialized radiologist by transvaginal and exclusive transuterine approach. Local anesthesia will be performed. A pain assessment will be performed during the biopsy (visual or verbal scale).

Between the biopsy and the procedure, the patient will be reviewed by the investigating surgeon to check the outcome of the biopsy, any pain or complications of the biopsy.

The surgical procedure will be performed by laparotomy and will consist of an extra-facial hysterectomy without fragmentation of the surgical specimen (extraction technique "in block"). During the procedure, the investigating surgeon will perform a description of the abdominal and pelvic cavity and perform a block excision of the tumor.

At one month of the surgery, patient will be reviewed by the investigating surgeon for a postoperative visit with clinical examination, gynecological and histopathological results.

Thereafter, the follow-up of the patients will be carried out according to the standards of care according to the histopathological results.

ELIGIBILITY:
Inclusion Criteria:

1. Woman >= 35 years old
2. Diagnosis of suspicious uterine tumor involving surgical management by laparoscopic hysterectomy with possible morcellation. Fibroma must be considered suspect, if at least one of the following characteristics is fulfilled:

   1. Rapid tumor growth defined as ≥30% of the maximum diameter in 1-year interval based on imaging findings, or,
   2. Symptomatic tumors in postmenopausal women presenting vaginal bleeding or pelvic pain or palpable masses or symptoms caused by pressure of neighbor organs such as dysuria and gastrointestinal symptoms, or,
   3. Tumors characterized by certain suspicious ultrasound criteria such as size > 8 cm, presence and distribution of vascularization, presence of intratumoral lesions, ultrasound heterogeneity, necrosis, cystic components, presence of calcification.
   4. Genetical predisposal to cancer syndromes such as Lynch syndrome, hereditary leiomyomatosis or "renal cell cancer".
3. MRI performed according to the technical and interpretation criteria stipulated in the study within 30 days before the biopsy.
4. Uterine fibroma accessible to transvaginal echo-guided biopsy exclusively.
5. No contraindication to performing laparotomy surgery.
6. Voluntary signed written informed consent.
7. Patient with a social security in compliance with the French law.

Exclusion Criteria:

1. General contraindication(s) to performing a transvaginal echo-guided biopsy.
2. Biopsy by peritoneal approach (surgical or percutaneous).
3. History of treated cancer in the two years preceding inclusion or in progressive continuation.
4. Unfavorable anesthetic assessment that does not allow general anesthesia for the planned surgery.
5. Coagulation disorders contraindicating biopsy.
6. Pregnancy project.
7. Pregnant or lactating woman.
8. Impossibility of submitting to the medical examination of the test for geographical, social or psychological reasons.
9. Patient deprived of liberty under legal protection measure or unable to express her consent.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity (Se) of preoperative vaginal ultrasound-guided biopsy (VUGB) in the pathological diagnosis of suspected sarcoma uterine tumors. | After surgery, an average of 2 months after inclusion
  Sensitivity is the proportion of patients with malignant/STUMP result on the local reading of biopsy (index test) divided by the number of patients with malignant/STUMP result on the local reading of surgical specimen (reference standard). Primary outcome assessment will be based on the local reading.

SECONDARY OUTCOMES:
Specificity (Sp) of VUGB in the pathological diagnosis of suspected sarcoma uterine tumors. | After surgery, an average of 2 months after inclusion
  Specificity is the proportion of patients with benign result on the local reading of biopsy divided by the number of patients with benign result on the local reading of surgical specimen.
Accuracy of VUGB in the pathological diagnosis of suspected sarcoma uterine tumors. | After surgery, an average of 2 months after inclusion
  Accuracy is the proportion of patients with true results: true positives (TP) + true negatives (TN) divided by number of cases. Accuracy ranges from 0 (100% false positives and false negatives) to 1 (100% true positives and true negatives). Assessment will be based on the local reading.
Youden's index (J) of VUGB in the pathological diagnosis of suspected sarcoma uterine tumors. | After surgery, an average of 2 months after inclusion
  Youden's index is defined as sensitivity+specificity-1. The maximum value of the Youden index is 1 (perfect test) and the minimum is 0 when the test has no diagnostic value. Assessment will be based on the local reading.
Positive Predictive Value (PPV) of VUGB in the pathological diagnosis of suspected sarcoma uterine tumors. | After surgery, an average of 2 months after inclusion
  PPV is the proportion of patients with malignant/STUMP results on the local reading of biopsy and surgical specimen (true positives) divided by the number of patients who might or might not have malignant/STUMP results (True positives+False positives).
Negative Predictive Value (NPV) of VUGB in the pathological diagnosis of suspected sarcoma uterine tumors. | After surgery, an average of 2 months after inclusion
  NPV is the proportion of patients with benign results on the local reading of biopsy and surgical specimen (true negatives) divided by the number of patients who might or might not have benign results (True negatives+ False negatives)
Sensitivity (Se) of preoperative vaginal ultrasound-guided biopsy (VUGB) in the pathological diagnosis of suspected sarcoma uterine tumors based on the centralized review by an expert pathologist. | After surgery, an average of 2 months after inclusion
  Sensitivity is the proportion of patients with malignant/STUMP result on the centralized review of biopsy (index test) divided by the number of patients with malignant/STUMP result on the centralized review of surgical specimen (reference standard).
Specificity (Sp) of VUGB in the pathological diagnosis of suspected sarcoma uterine tumors based on the centralized review by an expert pathologist. | After surgery, an average of 2 months after inclusion
  Specificity is the proportion of patients with benign result on the centralized review of biopsy divided by the number of patients with benign result on the centralized review of surgical specimen.
Accuracy of VUGB in the pathological diagnosis of suspected sarcoma uterine tumors based on the centralized review by an expert pathologist. | After surgery, an average of 2 months after inclusion
  Accuracy is the proportion of patients with true results: true positives (TP) + true negatives (TN) divided by number of cases. Accuracy ranges from 0 (100% false positives and false negatives) to 1 (100% true positives and true negatives). Assessment will be based on the centralized review by an expert pathologist.
Youden's index (J) of VUGB in the pathological diagnosis of suspected sarcoma uterine tumors based on the centralized review by an expert pathologist. | After surgery, an average of 2 months after inclusion
  Youden's index is defined as sensitivity+specificity-1. The maximum value of the Youden index is 1 (perfect test) and the minimum is 0 when the test has no diagnostic value. Assessment will be based on the centralized review by an expert pathologist.
Positive Predictive Value (PPV) of VUGB in the pathological diagnosis of suspected sarcoma uterine tumors based on the centralized review by an expert pathologist. | After surgery, an average of 2 months after inclusion
  PPV is the proportion of patients with malignant/STUMP results on the centralized review of biopsy and surgical specimen (true positives) divided by the number of patients who might or might not have malignant/STUMP results (True positives+False positives).
Negative Predictive Value (NPV) of VUGB in the pathological diagnosis of suspected sarcoma uterine tumors based on the centralized review by an expert pathologist. | After surgery, an average of 2 months after inclusion
  NPV is the proportion of patients with benign results on centralized review of biopsy and surgical specimen (true negatives) divided by the number of patients who might or might not have benign results (True negatives+ False negatives).
Sensitivity (Se) of imaging (MRI coupled with echo-guided biopsy) in the pathological diagnosis of suspected sarcoma uterine tumors. | After surgery, an average of 2 months after inclusion
  Sensitivity is the proportion of patients with malignant/STUMP result on imaging divided by the number of patients with malignant/STUMP result on the local reading of surgical specimen (reference standard).
Specificity (Sp) of imaging (MRI coupled with echo-guided biopsy) in the pathological diagnosis of suspected sarcoma uterine tumors. | After surgery, an average of 2 months after inclusion
  Specificity is the proportion of patients with benign result on imaging divided by the number of patients with benign result on the local reading of surgical specimen.
Accuracy of imaging (MRI coupled with echo-guided biopsy) in the pathological diagnosis of suspected sarcoma uterine tumors. | After surgery, an average of 2 months after inclusion
  Accuracy is the proportion of patients with true results: true positives (TP) + true negatives (TN) divided by number of cases. Accuracy ranges from 0 (100% false positives and false negatives) to 1 (100% true positives and true negatives).
Youden's index (J) of imaging (MRI coupled with echo-guided biopsy) in the pathological diagnosis of suspected sarcoma uterine tumors. | After surgery, an average of 2 months after inclusion
  Youden's index is defined as sensitivity+specificity-1. The maximum value of the Youden index is 1 (perfect test) and the minimum is 0 when the test has no diagnostic value.
Positive Predictive Value (PPV) of imaging (MRI coupled with echo-guided biopsy) in the pathological diagnosis of suspected sarcoma uterine tumors. | After surgery, an average of 2 months after inclusion
  PPV is the proportion of patients with malignant/STUMP results on imaging and surgical specimen (true positives) divided by the number of patients who might or might not have malignant/STUMP results (True positives+False positives).
Negative Predictive Value (NPV) of imaging (MRI coupled with echo-guided biopsy) in the pathological diagnosis of suspected sarcoma uterine tumors. | After surgery, an average of 2 months after inclusion
  NPV is the proportion of patients with benign results on Imaging and surgical specimen (true negatives) divided by the number of patients who might or might not have benign results (True negatives+ False negatives)
Reproducibility of local histopathological reading and centralized review by an expert pathologist of the echo-guided uterine biopsies. | After surgery, an average of 2 months after inclusion
  Cohen's Kappa coefficient. kappa coefficient values greater than 0.75 correspond to acceptable reproducibility.
Change From Baseline in Pain Scores on the Visual Analog Scale after biopsy. | at inclusion and after surgery (2 months after inclusion)
  The minimum value is 0 and the maximum value is 10. A high score of pain indicates a high level of pain.
Number of complications as assessed by the classification of Clavien-Dindo | After biopsy, an average of 1 day after inclusion.
  Complications related to biopsy will be evaluated after biopsy.
Number of adverse events as assessed by CTCAE v5.0 | an average of 2 months after inclusion
  Adverse events will be evaluated at inclusion, on the day of the biopsy and after the biopsy.
Progression-free survival (PFS) rate for atypical or dubious uterine sarcomas or fibroids (STUMP). | After surgery, an average of 3 years after surgery
  PFS is defined as the time interval between the date of surgery and the date of progression and/or death whichever occurs first
Overall survival (OS) rate for atypical or dubious uterine sarcomas or fibroids (STUMP). | After surgery, an average of 3 years after surgery
  OS is defined as the time interval between the date of surgery and the date of death (of any cause).

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric GUYON, Dr, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided